CLINICAL TRIAL: NCT04193865
Title: Hemofilter Life Span and Filtration of Inflammatory Markers in Patients Receiving Extracorporeal Life Support And/or Continuous Renal Replacement Therapy
Brief Title: Hemofilter Life Span, ECLS And/or CRRT
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 00094177
Record Dates: First submitted 2019-11-18; First posted 2019-12-10 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Kidney Diseases; Acute Injury of Kidney; Renal Failure; Renal Insufficiency; Neonatal Renal Disorder (Disorder)
Keywords: Extracorporeal life support; Extracorporeal membrane oxygenation; Acute Kidney Injury; Renal replacement therapy; Renal Support therapy; Kidney support therapy
MeSH Terms: conditions — Kidney Diseases; Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extracorporeal Life Support with Renal Replacement Therapy: This cohort will include all subjects receiving extracorporeal life support with concurrent continuous renal replacement therapy.
  Two blood samples and one ultrafiltration sample will be obtained for the study protocol twice per day (every 12 hours) for the duration of each participants's CRRT course.
- Renal Replacement Therapy: This cohort will include all subjects receiving continuous renal replacement therapy (no extracorporeal life support).
  Two blood samples and one ultrafiltration sample will be obtained for the study protocol twice per day (every 12 hours) for the duration of each patient's CRRT course.

SUMMARY:
The goal of this project to better understand the immune-modulatory effects of continuous renal replacement therapy (CRRT) in neonatal and pediatric patients, particularly those receiving extracorporeal life support (ECLS). Little is known about the effects of CRRT in this particular population and improved knowledge will be useful clinically and may lead to novel therapeutic approaches and improved outcomes for these critically ill patients.

DETAILED DESCRIPTION:
Via collection of serum and ultrafiltrate samples, the invesitgators will examine how hemofilter lifespan alters the filtration of pro- and anti-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal or pediatric patients receiving ECLS (>2 kilograms and >34 weeks gestation)
* CRRT utilized during ECLS course
* For the secondary endpoints comparing CRRT-mediated cytokine filtration in patients receiving ECLS with concurrent CRRT to patients receiving CRRT alone (no ECLS), the investigators will also enroll neonatal and pediatric patients receiving CRRT alone (no ECLS). Patients will be eligible for entry into this study if they meet all of the following criteria:
* Neonatal or pediatric patients receiving CRRT

Exclusion criteria:

-Those patients with inability or unwillingness of legal guardian/representative to give informed consent

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Both male and female neonatal (aged 0-28 days of life) and pediatric (children aged 29 days-17 years) patients receiving ECLS will be eligible. The study team will also enroll neonatal and pediatric patients receiving CRRT alone (no ECLS).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Cytokine concentrations over time (every 12 hours for the entire course of CRRT) | Cytokine concentrations over time every 12 hours for the entire course of CRRT through study completion, up to 12 months
  Quantify cytokine concentrations, specifically interferon (IFN)- γ, interleukin (IL)-1β, IL-6, IL-8, IL-10, IL-12p70, tumor necrosis factor (TNF)-α (all to result in concentrations in pg/ml), in pre-CRRT filter serum, post-CRRT filter serum, and ultrafiltrate (UF) using electrochemiluminescene assay and cytometric bead array and determine how age of the CRRT filter influences filtration of these cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Murphy, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No